Statistical analysis plan

Title Optimizing a self-directed mobile coping skills training

intervention to improve cardiorespiratory failure

survivors' psychological distress

Short title Blueprint

Principal Investigator(s) Christopher Cox

Co-Investigators Laura Porter, Sarah Kelleher

Biostatistician(s) Maren Olsen, Alice Parish

Version Date 10/22/21

IRB Pro00101848

ClinicalTrials.gov NCT04329702

10/22/21: SAP creation

**Activity Log** 

## 1 Study Overview

As survival has improved for the 2 million people with cardiorespiratory failure managed annually in US intensive care units (ICUs), it has become apparent that these patients suffer from severe and persistent post-discharge symptoms of psychological distress including depression, anxiety, and post-traumatic stress disorder (PTSD). However, few targeted interventions exist that are relevant to patients' experiences and that accommodate their many physical, social, and financial barriers to personalized care. To fill this gap, we have developed an innovative, native mobile coping skills training (CST) program that promotes automated care delivery and self-management of symptom-related distress. CST, by improving self-efficacy and adaptive coping, reduces psychological distress symptoms, thereby also improving quality of life.

Previous trials, in which this pilot randomized clinical trial (RCT) is based, have demonstrated that adaptive coping skills training (CST), is an active response for managing stressful events such as the experience of a critical illness. ICU survivors have emphasized in their own words the importance of coping to their perceived quality of life. While the use of adaptive coping skills (e.g., relaxation, positive reframing, problem solving) is associated with decreased psychological distress, ICU survivors infrequently apply such strategies.

This study is a 2 year pilot study that employs CST methods via a mobile app 'Blueprint'. There are 3 arms that participants can be randomized to: Intervention group 1 will receive access to the Blueprint app with a CST therapist introduction call (Arm 1), Intervention group 2 will receive access to the Blueprint app with no introduction call (Arm 2), or a control group of usual care with no access to the Blueprint app or introduction call (Arm 3). All participants will complete surveys at 4 timepoints: baseline (T0), discharge (T1), 1 month post discharge (T2), and 3 months post discharge (T3). The intervention groups will receive access to the Blueprint app which provides a 4 week course of various topics of CST skills. Participants in the intervention group are asked to utilize the app during their first month post-discharge.

## 1.1 Study Aims

#### 1.1.1 Primary Aim 1

Determine the feasibility and acceptability of the Blueprint app.

#### 1.1.2 Primary Aim 2

Determine the clinical impact on ICU survivors' 1 and 3 month psychological distress symptoms of intervention groups compared to usual care control.

## 1.2 Study Hypotheses

#### 1.2.1 Primary Hypothesis 1

The primary hypothesis is that the mobile CST app 'Blueprint' will be feasible and acceptable based on comparison of observed to a priori benchmarks.

#### 1.2.2 Primary Hypothesis 2

The secondary hypothesis is, compared to usual care, the intervention participants will have improvement in symptoms of psychological distress (HADS and PTSS scores) at the 1 and 3 month timepoints (T2 and T3).

## 2 Study Design and Study Population

Participants are patients who were admitted to the ICU and were critically ill with either respiratory failure/insufficiency or cardiac failure/insufficiency. Additionally, participants experienced a high level of distress (HADS  $\geq$ 8) at baseline.

This is a randomized clinical trial, where participants are consented and randomized to 1 of 3 arms (2 intervention arms, 1 control arm) in a 1:1:1 ratio. A total randomized sample size of 45 participants (15 per arm) was targeted. A method of minimization was used for randomization, with the aim to balance 3 stratification characteristics: ICU service (medical, surgical), baseline HADS score (<14,  $\ge14$ ), and age (<50,  $\ge50$ ).

#### 2.1 Inclusion Criteria

Patients included in Blueprint satisfied the following inclusion criteria:

At time of hospital admission:

- Age ≥ 18 years
- Managed in an adult ICU, step-down unit, <u>or</u> specialized care unit for ≥ 24 hours during the time in which inclusion criterion #3 is met.
- Presence of acute cardiac or respiratory failure, defined as having  $\geq 1$  of the following:
  - o Acute respiratory failure / insufficiency, defined as ≥1 of the following:
    - Mechanical ventilation via endotracheal tube for ≥4 hours
    - Non-invasive ventilation (CPAP, BiPAP) for ≥4 hours in a 24-hour period provided for acute respiratory failure in an ICU (not for obstructive sleep apnea or other stable use)
    - High flow / opti-flow nasal cannula or face mask oxygen use
    - ≥25% increase in baseline nasal cannula rate
  - o Acute cardiac failure / insufficiency, defined as ≥1 of the following:
    - use of vasopressors for shock of any etiology
    - use of inotropes for shock of any etiology
    - use of pulmonary vasodilators
    - use of aortic balloon pump or cardiac assist device for cardiogenic shock
    - use of diuretic intravenous drip
- Cognitive status intact, defined as:
  - No history of significant cognitive impairment (e.g., dementia)
  - Absence of current, significant cognitive impairment (≥ 3 errors on the Callahan cognitive status screen)
  - Decisional capacity present
- Absence of severe and/or persistent serious mental illness that could disrupt study participation, as noted in the electronic medical record (EMR) or affirmed by clinical staff at the time of screening and approach for consent. Defined as any of the following:

- o Treatment for severe or unstable mental illness (e.g., psychosis, schizophrenia) within the last 6 months preceding the current hospital admission
- o Active substance abuse that impairs ability to participate
- o Endorsing suicidality at time of admission or informed consent discussion
- English fluency.

#### At time of discharge:

• Elevated baseline psychological distress symptoms, defined as HADS total score of  $\geq 8$  at the completion of survey 1, T1.

#### 2.2 Exclusion Criteria

Patients were excluded from Blueprint if they satisfied the following exclusion criteria:

At time of hospital admission:

- Complex medical care expected soon after discharge (e.g., planned surgeries, transplantation evaluation, extensive travel needs for follow up care, disruptive chemotherapy/radiation regimen)
- Unable to complete study procedures as determined by staff.
- Lack of access to either reliable smartphone with cellular data plan or wifi

At time of hospital discharge:

- Failure to randomize within 1 month after discharge from the hospital to home.
- Failure to access app within 1 month after randomization.

The following additional exclusion criteria were applied after data collection:

• Any data recorded after a participant has withdrawn

## 2.3 Data Acquisition

 $File \ path \ for \ raw\ data: .. \ \ CRU \ Pulmonary \ Christopher\ Cox \ Pro00101848\ mCST\ Blueprint \ Main\ Analysis \ DATA \ RAW$ 

| File Name | Description |
|---------------------------------|---------------------------------------|
| Blueprint Data Export XXXX.xlsx | Blueprint App data pulled by Jennifer |
| | This file has multiple sheets. |
| BlueprintScreeningAn_SAS_xxxx | Blueprint REDCap data pulled by Alice |

Note: Data will be analyzed in SAS 9.4.

## 3 Outcomes, Exposures, and Variables of Interest

## 3.1 Primary Outcome(s)

| Variable | Dataset | Description | Specifications |
|----------|---------|-------------|----------------|

| hads | Blueprint/Baseline | HADS total score<br>at T0 | Continuous |
|---|---|---|---|
| Hads | Blueprint/T1 | HADS total score<br>at T1 | Continuous (may need to be derived from item scores HADS01—HADS14) |
| Score_hads | Blueprint/T2 | HADS total score<br>at T2 | Continuous (may need to be derived from item scores HADS01—HADS14) |
| Score_hads | Blueprint/T3 | HADS total score<br>at T3 | Continuous (may need to be derived from item scores HADS01—HADS14) |
| ptss | Blueprint/T1 | PTSS total score<br>at T1 | Continuous (may need to be derived from item scores ptss_1— ptss_10) |
| Score_ptss | Blueprint/T2 | PTSS total score<br>at T2 | Continuous (may need to be derived from item scores ptss_1— ptss_10) |
| Score_ptss | Blueprint/T3 | PTSS total score<br>at T3 | Continuous (may need to be derived from item scores ptss_1— ptss_10) |
| D3mo_HADS | Blueprint/T3<br>Blueprint/T1 | Change in HADS at 3 months | Derived as Score_hads(T3) - ??? |
| D1mo_HADS | Blueprint/T2<br>Blueprint/T1 | Change in HADS at 1 months | Derived as Score_hads(T2) - ??? |
| D3mo_PTSS | Blueprint/T3<br>Blueprint/T1 | Change in PTSS at 3 months | Derived as Score_ptss(T3) - ??? |
| D1mo_PTSS | Blueprint/T2<br>Blueprint/T1 | Change in PTSS at 1 months | Derived as Score_ptss(T2) - ??? |
| ADLs/IADLs | T1, t2, t3 | | Not really an outcome but |
| Systems Usability<br>Scale | T1 | | |
| PHQ-10 physical symptom scale | T1, t2, t3 | | |
| Quality of life 100-<br>point VAS | T1, t2, t3 | | |
| List | | Feasibility | Eligibility: 70% of positive screens Consent: 80% of eligible Randomized: 80% of consented Retention: 80% Adherence: 75% of tasks ***note that these need to be defined a bit more specifically |
| CSQ-8 | ` | Acceptability | |

## 3.2 Primary Exposure(s)

| Variable | Dataset | Description | Specifications |
|---|---|---|---|
| Plan_name | Blueprint/Participants | Trial Arm | A multi-level categorical variable |
| | | | - Blueprint Screening & Baseline: |
| | | | Exclude |
| | | | - Blueprint (Group 1): Arm 1 |
| | | | - Blueprint (Group 2): Arm 2 |
| | | | - Blueprint (Control): Arm 3 |

#### 3.3 Other Variables of interest

| Variable | Dataset | Description | Specifications |
|----------|---------|-------------|----------------|

## 4 Statistical Analysis Plan

All analyses will be done using SAS 9.4. Continuous variables will be summarized with mean/standard deviation/median/Q1-Q3/range and categorical variables with frequency counts and percentages. Number of missing data for each variable will be reported.

## 4.1 Analysis Plan for Primary Aim 1

- 1. First, we will describe our cohort. In Table 1 we will summarize participant characteristics overall and by arm. No statistical tests will be provided as this was a randomized trial, and ideally groups should be balanced.
- 2. To assess Aim 1 for feasibility and acceptability we will evaluate CSQ-8 and SUS scores. Results will be reported in Table 2.

## 4.2 Analysis Plan for Primary Aim 2

- 1. To address Aim 2, we will describe the secondary outcomes at each time point by arm, as well as the change in scores at T2 and T3 from T1 in Table 3. Any additional secondary outcomes will be described in this table.
- 2. To assess if there was change at each timepoint of interest between the arms we estimate mean changes (and 95% CI) from baseline to each timepoint for each distress outcome (HADS, PTSS) using a general linear model (PROC MIXED). Model parameters will include treatment arm (1, 2, 3), time indicator (T1, T2, T3), and an arm by time interaction term. Change estimates and CI's will be reported in Table 4. To quantify clinically important differences, rather than report p-values which is not recommended for pilot studies with

small sample sizes, we will compare the estimated group mean differences and 95% CI's to half (0.5) of the baseline standard deviation (SD) of each outcome score.

# 5 Appendix I: Planned figures and tables

Figure 1: CONSORT Diagram

Table 1: Demographic characteristics of participants at baseline

| Characteristic | Group 1 | Arm 2:<br>Intervention<br>Group 2<br>(Blueprint<br>only)<br>N= | Control | Total<br>N= |
|---|---|---|---|---|
| Stratification Variables | | | | |
| Age | | | | |
| <50 | | | | |
| ≥50 | | | | |
| ICU Service | | | | |
| Medical | | | | |
| Surgical | | | | |
| Baseline HADS | | | | |
| <14 | | | | |
| ≥14 | | | | |
| Other Baseline Characteristics | | | | |
| Age | | | | |
| Mean (sd) | | | | |
| Median | | | | |
| Q1, Q3 | | | | |
| Range | | | | |
| Gender | | | | |
| Male | | | | |
| Female | | | | |

Table 2: Feasibility and Acceptability

| Characteristic | Arm 1: Arm 2: Intervention Intervention | Arm 3:<br>Control | Total |
|---|---|---|---|
| | Group 1 | (Usual Care) | N= |

| | (Blueprint +<br>Therapist)<br>N= | • | N= |
|------------------------------|----------------------------------|---|----|
| Feasibility | | | |
| % Consented | | | |
| % Randomized | | | |
| % Retained | | | |
| % Completed Surveys | | | |
| T1 | | | |
| T2 | | | |
| T3 | | | |
| All timepoints | | | |
| % Completed all intervention | | | |
| components | | | |
| Acceptability | | | |
| CSQ Score | | | |

 Table 3: Participant Outcomes

| Characteristic | Arm 1:<br>Intervention<br>Group 1<br>(Blueprint +<br>Therapist)<br>N= | Arm 2:<br>Intervention<br>Group 2<br>(Blueprint<br>only)<br>N= | Arm 3:<br>Control<br>(Usual Care)<br>N= | Total<br>N= |
|---|---|---|---|---|
| Hospital LOS (Discharge – admission) | | | | |
| Hospital discharge disposition | | | | |
| 3 month disposition | | | | |

**Table 4:** Observed and Estimated mean score and differences by Arm and Time for HADS and PTSS outcomes

| | Baseline | 1 Month | 3 Months | Δ1 month - | Δ3 months- |
|---|---|---|---|---|---|
| | (T1?) | (T2) | (T3) | Baseline | Baseline |
| HADS | | | | | |
| Observed Score | | | | | |
| Arm 1 (BP + | | | | | |
| Therapist) | | | | | |
| Arm 2 (BP only) | | | | | |
| Arm 3 (Control) | | | | | |
| <b>Estimated Mean S</b> | Estimated Mean Score (95% CI) | | | | |
| Arm 1 (BP + | | | | | |
| Therapist) | | | | | |
| Arm 2 (BP only) | | | | | |

| Arm 3 (Control) | |
|-------------------------|---------------|
| Diff (Arm 1 - | |
| Arm 3) | |
| Diff (Arm 2 – | |
| Arm 3) | |
| PTSS | |
| Observed Score | |
| Arm 1 (BP + | |
| Therapist) | |
| Arm 2 (BP only) | |
| Arm 3 (Control) | |
| <b>Estimated Mean S</b> | core (95% CI) |
| Arm 1 (BP + | |
| Therapist) | |
| Arm 2 (BP only) | |
| Arm 3 (Control) | |
| Diff (Arm 1 - | |
| Arm 3) | |
| Diff (Arm 2 - | |
| Arm 3) | |